CLINICAL TRIAL: NCT06675864
Title: An Open-label, Multi-center, Phase I/II Study to Assess Safety, Disease Progression, and Cellular Kinetics Following YTB323 Administration in Participants With Non-active Progressive Multiple Sclerosis (PMS)
Brief Title: Open-label, Multi-center, Phase I/II Study to Assess Safety, Disease Progression and Cellular Kinetics Following YTB323 Administration in Participants With Non-active Progressive Multiple Sclerosis (PMS)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYTB323r12101
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Chimeric Antigen Receptor T cells; CAR-T; YTB323; Multiple Sclerosis; MS; Progressive Multiple Sclerosis; PMS; rapcabtagene autoleucel
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- YTB323 Cohort 1 (Experimental): Participants will receive one dose of YTB323
  Interventions: Biological: rapcabtagene autoleucel (YTB323)
- YTB323 Cohort 2 (Experimental): Participants will receive one dose of YTB323
  Interventions: Biological: rapcabtagene autoleucel (YTB323)
- YTB323 Cohort 3 (Experimental): Participants will receive one dose of YTB323
  Interventions: Biological: rapcabtagene autoleucel (YTB323)
- YTB323 Cohort 4 (Experimental): Participants will receive one dose of YTB323
  Interventions: Biological: rapcabtagene autoleucel (YTB323)

INTERVENTIONS:
Biological: rapcabtagene autoleucel (YTB323) — CAR-T cell suspension for intravenous infusion

SUMMARY:
This is an open-label, multi-center, non-confirmatory study to assess the safety, disease progression, and cellular kinetics following YTB323 administration to 28 participants with non-active Progressive Multiple Sclerosis (PMS). The study design utilizes an ascending single dose design consisting of 3 sentinel cohorts followed by an expansion cohort.

DETAILED DESCRIPTION:
All participants in this study will receive YTB323. Both the participant and the study doctor will know the participant is getting YTB323. Participants will be given one dose of YTB323. Different groups of participants may receive a higher dose of YTB323, if proven to be safe for every participant at the lower dose. Participants are in this study for 2 years and will be followed for an additional 13 years in a long-term follow up study. The main question this trial is designed to answer: Is YTB323 treatment safe for participants with progressive MS?

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female participants 18 to 60 years (inclusive) at screening.
2. Signed informed consent must be obtained prior to participation in the study.
3. Able to communicate well with the investigator, to understand and comply with the requirements of the study including:

   * Able to undergo lumbar puncture (LP), blood draws, tolerate brain and spinal MRI, and able to participate and tolerate all study procedures at study visits.
4. Diagnosis of SPMS or PPMS according to the 2017 McDonald diagnostic criteria (Thompson et al 2018) as confirmed at screening visit.
5. Less than 15 years (inclusive) from onset of first MS symptoms as determined by the investigator during screening.
6. Ambulatory Patients (EDSS 3 to 6.5 inclusive) at screening.
7. Evidence of recent (within 24 months) disease progression of ≥1.00 on the EDSS scale.
8. No relapse in the last 24 months at screening.
9. No Gd-enhancing lesion on brain or spinal cord MRI at screening.
10. Participants must receive or be current on all recommended vaccinations according to institutional, local, or global guidelines for immunocompromised patients at least 6 weeks prior to lymphodepletion.

Key Exclusion Criteria:

1. Diagnosis of relapsing multiple sclerosis (RMS) or active PMS according to the 2017 revision of the McDonald diagnostic criteria (Thompson et al 2018) at screening.
2. History of, or current, clinically significant CNS disease except MS (e.g. stroke, traumatic brain or spinal injury, history or presence of myelopathy, history of seizures or epilepsy) or neurological disorders which may mimic MS at screening.
3. Evidence of clinically significant cardiovascular (such as but not limited to myocardial infarction, unstable ischemic heart disease, New York Heart Association Class III/IV left ventricular failure, arrhythmia and uncontrolled hypertension within 6 months prior to or during screening).
4. Participants with history of confirmed Progressive Multifocal Leukoencephalopathy (PML) or neurological symptoms consistent with PML prior to or during screening.
5. Clinically significant, active, opportunistic, chronic or recurrent infection (including positive for hepatitis B or hepatitis C) confirmed by clinical evidence, imaging, or positive laboratory tests one month prior to leukapheresis.
6. Have donated blood or experienced a loss of blood > 400 mL within 3 months prior screening, or longer if required by local regulations.
7. Any prior stem cell therapy or organ transplantation or gene therapy.
8. Any contraindications to LP, including but not limited to:

   * Known or suspected structural abnormality of the lumbar spine that, in the opinion of the Investigator, may interfere with the performance of the LP, or increase the risk of the procedure for the participant.
   * Presence of risk for increased or uncontrolled bleeding (including but not limited to vascular abnormalities or neoplasms at or near the LP site, disorders of the coagulation cascade, platelet function, or platelet count).
   * Participants on anticoagulants (e.g., warfarin) or antiplatelets [except for low-dose aspirin (100 mg/day or lower) and low-dose nonsteroidal anti-inflammatory drugs such as ibuprofen (600 mg/day or lower) which are allowed], are not eligible to participate.
9. Not willing or able to have MRI scans as per protocol e.g. due to claustrophobia, or absolute contraindications to MRI (e.g., metallic implants, metallic foreign bodies, pacemaker, defibrillator).
10. Pregnant or nursing (lactating) women.
11. Past surgical history of splenectomy.
12. Evidence of active or latent tuberculosis (TB) infection by QuantiFERON® TB-Gold assay (or equivalent) performed at Screening by central lab. In case of unclear or indeterminate test results, the Investigator should consult with an infectious disease expert to exclude the diagnosis of active or latent TB infection and document this in the source data. Participant should be excluded if they have any signs of active TB observed in available lung imaging (e.g., X-ray or HRCT).
13. Any psychiatric, pulmonary (including, history of or active severe respiratory disease, including Chronic Obstructive Pulmonary Disease, interstitial lung disease or pulmonary fibrosis), renal, hepatic, endocrine, metabolic (e.g. severe hypoproteinemia due to nephrotic syndrome), hematological disorders or gastrointestinal disease that, in the investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the participant, prior to or during screening.
14. Grade 2 or higher thromboembolic event in the past 4 weeks prior to or during Screening or evidence of disorders of coagulation or platelet function including subjects that require chronic use of anticoagulation or antiplatelet drugs (please refer to the key exclusion criteria no. 8 for the exceptions).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2030-06-14 (Estimated); Study Completion 2030-06-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs), Adverse Events (AEs), and Serious Adverse Events (SAEs) | Day 1 through Year 2
  Occurrence, severity, and frequency of dose limiting toxicities (DLTs), AEs and SAEs, including changes in vital signs, electrocardiograms (ECGs), laboratory parameters, neurological status and magnetic resonance (MRI) of the brain and spinal cord qualifying and reported as AEs.

SECONDARY OUTCOMES:
Measure of Disability: Expanded Disability Status Scale (EDSS). | Day 1 through Year 2
  EDSS is used to measure the change in disability level in participants using a scale from 0 to 10. The higher the score, the greater the degree of disability.
Measure of Disability: Short Form Health Survey (SF-36 v2) | Day 1 through Year 2
  The Short Form Health Survey (SF-36 v2) is a widely used and extensively studied instrument to measure health-related quality of life among healthy participants and participants with acute and chronic conditions. It consists of eight subscales that can be scored individually: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. Two overall summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS) also can be computed. The SF 36 has proven useful in monitoring general and specific populations, comparing the relative burden of different diseases, differentiating the health benefits produced by different treatments, and in screening individual participants.
Measure of Disability: Timed 25 Foot Walk (T25FW) | Day 1 through Year 2
  The T25FW is a mobility test based on a timed walk of 25 feet that is administered by a trained administrator. The participant is directed to walk the clearly marked 25-foot distance as quickly as possible. Longer completion time corresponds with decreased mobility.
Measure of Disability: 9 Hole Peg Test (9HPT) | Day 1 through Year 2
  The 9HPT is a finger dexterity test that is administered by a trained administrator. The participant is directed to put 9 pegs, one by one, onto and then off the holder board as quickly as possible starting with using only the dominant hand, and then repeated with the non-dominant hand. Longer completion times are associated with decreased finger dexterity.
Measure of Disability: Symbol Digit Modalities Test (SDMT) | Day 1 through Year 2
  The SDMT is a timed cognition test administered by a trained administrator. The test assesses sustained attention, processing speed, visual scanning, and motor speed to determine cognitive impairment. Participants are given a coding key which contains abstract symbols that correspond to specific numbers. Participants are timed how quickly and accurately they are able to substitute the symbols for the numbers and is scored by the number of correctly coded items.
Modified Fatigue Impact Scale (MFIS) | Day 1 through Year 2
  The MFIS is a questionnaire to assess fatigue-related symptoms in patients with MS.
Whole Blood Pharmacokinetics (PK) of YTB323 - CMAX | Day 1 through Year 2
  Measured by Cmax - The maximum plasma concentration of YTB323
Whole Blood Pharmacokinetics (PK) of YTB323 - AUC | Day 1 Through Year 2
  Measured by AUC - Area under the curve of YTB323
Whole Blood Pharmacokinetics (PK) of YTB323 - Tmax | Day 1 Through Year 2
  Measured by Tmax - Time to Reach the Maximum Concentration After Drug Administration of YTB323
Whole Blood Pharmacokinetics (PK) of YTB323 - Clast | Day 1 Through Year 2
  Clast is defined as the Last observed (quantifiable) plasma concentration (Clast
Whole Blood Pharmacokinetics (PK) of YTB323 - Tlast | Day 1 through Year 2
  Tlast is defined as Time of Last Measurable Concentration
Humoral Immunogenicity of YTB323 | Day 1 through Year 2
  Incidence and prevalence of pre-existing and treatment induced humoral immunogenicity of YTB323
Cellular Immunogenicity of YTB323 | Day 1 through Year 2
  Incidence and prevalence of pre-existing and treatment induced cellular immunogenicity of YTB323
Safety data including dose limiting toxicities (DLTs), Adverse Events (AEs), and Serious Adverse Events (SAEs) from each dose level | Day 1 through Year 2
  Safety data from each dose level will be used to assess safe dose-level(s) to be continued in phase 2 and later clinical studies

CONTACTS AND LOCATIONS:
Locations (17):
- Australia (2):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
- Novartis Investigative Site, Québec, Quebec, Canada
- France (4):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Rennes
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Ulm
- Italy (2):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Málaga
- Switzerland (3):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com